CLINICAL TRIAL: NCT06331195
Title: Effects of an Adapted Brazilian Cardioprotective Diet Supplemented or Not With Phytosterols and/or Krill Oil in Patients With Familial Hypercholesterolemia: the DICA-FH Randomized Clinical Trial
Brief Title: An Adapted Brazilian Cardioprotective Diet, Phytosterols and Krill Oil in Familial Hypercholesterolemia (DICA-FH)
Acronym: DICA-FH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DICA-HF_MAIN
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DICA-FH + placebo (Placebo Comparator): Participants allocated into this arm (n= 75) will receive the DICA Br adapted to FH (DICA-FH) plus placebo of both phytosterol and krill oil during 120 days.
  Interventions: Other: Placebo phytosterol; Other: Placebo krill oil
- DICA-FH + phytosterol (Experimental): Participants allocated into this arm (n= 75) will receive the DICA Br adapted to FH (DICA-FH) plus 2g/day of phytosterol and placebo of the krill oil during 120 days.
  Interventions: Other: Placebo krill oil; Dietary Supplement: Phytosterol
- DICA-HF + krill oil (Experimental): Participants allocated into this arm (n= 75) will receive the DICA Br adapted to FH (DICA-FH) plus 2g/day of krill oil and placebo of phytosterol during 120 days.
  Interventions: Other: Placebo phytosterol; Dietary Supplement: Krill oil
- DICA-HF + phytosterol + krill oil (Experimental): Participants allocated into this arm (n= 75) will receive the DICA Br adapted to FH (DICA-FH) plus 2g/day of phytosterol and 2g/day of krill oil during 120 days.
  Interventions: Dietary Supplement: Phytosterol; Dietary Supplement: Krill oil

INTERVENTIONS:
Other: Placebo phytosterol — Placebo of phytosterol, in the same quantity of the active phytosterol.
  Arms: DICA-FH + placebo; DICA-HF + krill oil
Other: Placebo krill oil — Placebo of krill oil, in the same quantity of the active krill oil.
  Arms: DICA-FH + phytosterol; DICA-FH + placebo
Dietary Supplement: Phytosterol — 2g/day will be provided to the participants, aiming to guarantee a minimum of 800mg/day of free phytosterols.
  Arms: DICA-FH + phytosterol; DICA-HF + phytosterol + krill oil
Dietary Supplement: Krill oil — 2g/day will be provided to the participants, aiming to guarantee a minimum of 400mg/day of eicosapentaenoic (EPA) and docosahexaenoic (DHA) fatty acids.
  Arms: DICA-HF + krill oil; DICA-HF + phytosterol + krill oil

SUMMARY:
The main objective of this randomized clinical trial is to evaluate the effects of the adapted Brazilian Cardioprotective Diet (DICA Br) supplemented or not with phytosterols and/or krill oil in patients with a probable or definitive diagnosis of familial hypercholesterolemia (FH) according to the the Dutch Lipid Clinic Network (Dutch MEDPED) criteria. In addition, the following will be considered secondary objectives: to perform participants´ whole genome sequencing (WGS); to evaluate the effects of the interventions on lipid profile biomarkers; to evaluate the frequency of mild, moderate and severe adverse events according to study groups; and to evaluate adherence rates according to study groups. In this study, 300 individuals will be randomly enrolled into four groups: 1) DICA Br adapted to the FH context (DICA-FH) + phytosterol placebo + krill oil placebo (control group); 2) DICA-FH + 2g/day of phytosterol + krill oil placebo; 3) DICA-FH + phytosterol placebo + 2g/day of krill oil; and 4) DICA-FH + 2g/day of phytosterol + 2g/day of krill oil. Primary outcomes will be LDL-cholesterol for groups phytosterol vs. placebo and lipoprotein(a) for groups krill oil vs. placebo after 120 days of follow up.

DETAILED DESCRIPTION:
DICA-FH study is a superiority, factorial, and in parallel multicenter randomized placebo-controlled (double-dummy) clinical trial. The randomization will be in blocks stratified by research center, and the allocation ratio will be 1:1:1:1. Participants will come from at least 20 center sites in different Brazilian geographic regions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years;
* Definitive (certainty) or probable diagnosis of FH by the Dutch MEDPED criteria;
* Using one of the following treatment regimens for ≥6 weeks according to age:

>= 20 years -> simvastatin 40 mg; lovastatin 40 mg; pravastatin 80 mg; atorvastatin 20 mg; rosuvastatin 10 mg; pitavastatin 4 mg; fluvastatin 80 mg; atorvastatin 40- 80 mg; rosuvastatin 20 - 40 mg; atorvastatin 40 - 80 mg + ezetimibe 10mg; rosuvastatin 20 - 40 mg + ezetimibe 10mg; or simvastatin 40mg + ezetimibe 10mg.

16 to 19 years -> simvastatin 10 - 40 mg; lovastatin 10 - 40 mg; pravastatin 10 - 40 mg; atorvastatin 10 - 40 mg; rosuvastatin 5 - 40 mg; cholestyramine 4 to 16 mg; ezetimibe 10mg (in combination with statin).

Exclusion Criteria:

* Having a "possible" FH result according to the Dutch MEDPED criteria;
* TG ≥ 500mg/dL up to 6 months before screening for the study;
* Diagnosis of hypercholesterolemia due to a secondary cause recorded in the medical record;
* Food allergies (foods, dyes, preservatives);
* Contraindication to the use of phytosterols (for example: diagnosis of sitosterolemia);
* HIV positive on treatment with detectable viral load or AIDS;
* Chronic inflammatory or autoimmune diseases;
* Known liver disease, chronic kidney disease on dialysis or pancreatitis (acute and chronic);
* Cancer being treated or life expectancy < 6 months;
* Episode of acute coronary syndrome in the last 60 days;
* Chemical dependency/alcoholism;
* Chronic use of anti-inflammatories, anticonvulsants and immunosuppressive drugs;
* Use of PCSK9 inhibitors (alirocumab, evolocumab, inclisiran);
* Pregnancy or lactation;
* Individuals who are unable to perform an anthropometric assessment, at the discretion of the investigator;
* Grade III/severe obesity (body mass index [BMI] ≥40kg/m² for adults or percentile >99.9 or z-score >+3 according to WHO/2006 growth curves for BMI/Age indicator for adolescents);
* Use of dietary supplements that may interfere with the outcomes of interest (dietary fiber modules, n-3 PUFA, essential fatty acids);
* Participation in other randomized clinical trials;
* Refusal to participate in the study, due to failure to sign the Free and Informed Consent Form.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
LDL-c | 120 days
  Low-density lipoprotein cholesterol, in mg/dL
Lp(a) | 120 days
  Lipoprotein(a), in mg/dL

SECONDARY OUTCOMES:
TC | 120 days
  Total cholesterol, in mg/dL
HDL-c | 120 days
  High density lipoprotein cholesterol, in mg/dL
TG | 120 days
  Fasting triglycerides, in mg/dL
VLDL | 120 days
  Very low-density lipoprotein cholesterol, in mg/dL
NHDL | 120 days
  Non-HDL cholesterol, in mg/dL, calculated according to the mathematical formula: CT - HDL-c
CI I | 120 days
  Castelli Index I, in mg/dL, calculated according to the mathematical formula: CT/HDL-c
CI II | 120 days
  Castelli Index II, in mg/dL, calculated according to the mathematical formula: LDL-c/HDL-c
TG/HDL-c | 120 days
  TG/HDL-c ratio, in mg/dL, calculated according to the mathematical formula: TG/HDL-c TG/HDL-c ratio, in mg/dL, calculated according to the mathematical formula: TG/HDL-c
AI | 120 days
  Atherogenic index, in mg/dL, calculated according to the mathematical formula: NHDL/HDL-c
ox-LDL | 120 days
  Oxidized LDL, in µg/mL
APOAI | 120 days
  Apolipoprotein A-I, in mg/dL
APOB100 | 120 days
  Apolipoprotein B-100, in mg/dL
AE | 120 days
  Adverse events (mild, moderate and severe), registered as percentage per study group
Adherence | 120 days
  Adherence to treatment, evaluated by: attendance at consultations (at least 3 of the 4 planned study visits); diet quality; plasma concentrations of phytosterols and erythrocyte levels of EPA/DHA fatty acids (identified by the difference between the last and the first study visits); and counting the consumed products under investigation (consumption of at least 80% of the capsules provided to the participants, regardless of the allocation group).

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Hospital do Coracao; Rachel Helena Machado, MSc, Study Chair — Hospital do Coracao; Erlon O Abreu-Silva, MSc, Study Chair — Hospital do Coracao
Locations (24):
- Brazil (24):
  - Hcor, São Paulo, São Paulo
  - OCARA, Belém
  - Centro Oncológico de Roraima, Boa Vista
  - Instituto de Cardiologia e Transplantes do DF, Brasília
  - Universidade do Mato Grosso do Sul, Campo Grande
  - Universidade Federal do Mato Grosso, Cuiabá
  - Hospital Oto Aldeota, Fortaleza
  - Universidade Federal de Goiás, Goiânia
  - Universidade Federal do Amapá, Macapá
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió
  - Universidade Federal do Amazonas, Manaus
  - Universidade Estadual de Maringá, Maringá
  - Santa Casa de Montes Claros, Montes Claros
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas, Natal
  - Universidade Federal do Tocantins, Palmas
  - Universidade Federal do Vale do São Francisco, Petrolina
  - Instituto de Pesquisa e Ensino em Saúde, Porto Velho
  - Centro de Pesquisa Silvestre Santé, Rio Branco
  - Instituto Nacional de Cardiologia, Rio de Janeiro
  - Hospital Ana Nery, Salvador
  - InCor, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Universidade Federal de São Paulo, São Paulo
  - Centro de Pesquisa Cardiolima, Teresina

IPD SHARING:
Plan to Share IPD: Undecided